CLINICAL TRIAL: NCT02357121
Title: Focal Laser Ablation of Prostate Tissue: A Pilot Feasibility Study Using MRI/US Image Fusion for Guidance
Brief Title: Focal Laser Ablation of Prostate Tissue
Acronym: FLA
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Jean Perkins Foundation (Unknown); Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-000018; JCCCID534 (Other: Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2015-01-28; First posted 2015-02-06 (Estimated); Last update posted 2020-09-21 (Actual); Status verified 2020-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Laser ablation (Experimental): All patient will undergo focal ablation of prostate tissue utilizing laser energy.
  Interventions: Device: Focal Laser Ablation

INTERVENTIONS:
Device: Focal Laser Ablation — Focal laser ablation of prostate tissue using laser interstitial thermal therapy (LITT) under MR/ultrasound fusion guidance
  Other Names: laser treatment

SUMMARY:
This is an open-label pilot, feasibility/exploratory study to evaluate the safety of laser interstitial thermal therapy (LITT) using Visualase in the focal ablation of prostate tissue and to gather data for the design of future studies. Intra-procedure temperature and concurrent rectal wall thermistor monitoring will be performed for internal validation. Subjects will be monitored for adverse events, and health-related quality of life (HRQOL) questionnaires will be obtained. Post-treatment MRI and biopsies will be obtained to evaluate histologic and radiologic changes. Biomarker (PSA, PCA3 and PHI) kinetics will also be monitored.

ELIGIBILITY:
Inclusion Criteria

* Subjects with untreated organ confined prostate cancer (clinical stage ≤ T2b, Gleason ≤ 3+4)
* Negative metastatic workup with bone scan and CT abdomen/pelvis, within 6 months of study treatment, if indicated by PSA >10
* Age 40 years to 85 years of age
* Multi-parametric MRI at UCLA within 6 months of study treatment, demonstrating a

  * Region of interest (ROI) of MRI suspicion level 3 or higher
  * MRI-calculated prostate volume 25cc to 100cc
* Transrectal ultrasound-guided biopsy with ≥ 10 systematic biopsy cores and ≥ 2 MRI-ultrasound fusion targeted biopsy cores from above MRI-derived ROI

  * Histologically-confirmed adenocarcinoma from targeted biopsy cores
  * Overall Gleason score not to exceed 3+4
* Subjects desire focal therapy and decline conventional treatment (active surveillance, radical prostatectomy, radiation therapy, cryosurgery and hormone therapy)
* Signed informed consent for the FLA treatment through the 12 month follow up visit.

Exclusion Criteria:

* Any significant cancer outside of MRI target (ROI) area, defined as Gleason score > 3+4

  * < 10 years life expectancy
  * American Society of Anesthesiologists (ASA) criteria of IV or higher
  * Unfit for conscious sedation anesthesia
  * Active bleeding disorder as determined by abnormal prothrombin time, partial thromboplastin time, INR or platelet count (as determined by institutional lab parameters) at the time of screening
  * Use of coumadin or any other anticoagulant, unless anticoagulation can be temporarily reversed or stopped for a window of at least 7 days peri-procedure
  * Active urinary tract infection
  * Prostate abscess, chronic or acute prostatitis, or neurogenic bladder
  * Any prior treatment for prostate cancer

    * Radical prostatectomy
    * Radiation therapy (external beam or brachytherapy)
    * Cryotherapy
    * High intensity focused ultrasound treatment
    * Photodynamic therapy
    * Androgen deprivation therapy
  * Prior prostate, bladder neck, or urethral stricture surgery

    * Any prostate debulking procedure, including: transurethral resection of prostate, photovaporization, or electrovaporization
    * Transurethral incision of bladder neck
    * Urethral stricture dilation or reconstruction
  * Any current 5-alpha reductase inhibitors (history of use ≥ 3 months prior to MRI is acceptable)
  * Prior significant rectal surgery (hemorrhoidectomy is acceptable)
  * Rectal fissure, fibrosis, stenosis, or other anatomic abnormality precluding insertion of transrectal device
  * Inflammatory bowel disease
  * Urinary tract or rectal fistula
  * Any contraindication to MRI (contrast allergy severe claustrophobia, MRI-incompatible prosthesis)

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-09-17 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
safety of focal laser treatment using LITT: Number of participants with adverse events | 12 months
  Number of participants with adverse events will be collected in the 12 month follow-up period to assess safety.

SECONDARY OUTCOMES:
Efficacy of focal laser ablation of prostate tissue using the LITT system. | 12 months
  MRI changes will be determined at 6 and 12 months post FLA to assess efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Marks, MD, Principal Investigator — University of California at Los Angeles
Locations (2):
- United States (2):
  - UCLA, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California